CLINICAL TRIAL: NCT00400400
Title: A 4-week, Multicenter, Double-blind, Double-dummy, Randomized, Parallel Group Study to Compare the Gastrointestinal Safety and Tolerability of EC-MPS & MMF When Administered in Combination With Calcineurin Inhibitors in Renal Transplant Recipients Experiencing Gastrointestinal Intolerance
Brief Title: Enteric-coated Mycophenolate Sodium (EC-MPS) and Mycophenolate Mofetil (MMF) in Renal Transplant Patients With Gastrointestinal (GI) Intolerance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CERL080AUS51
Record Dates: First submitted 2006-11-15; First posted 2006-11-16 (Estimated); Results first posted 2011-08-15 (Estimated); Last update posted 2011-08-15 (Estimated); Status verified 2011-07

CONDITIONS: Renal Transplantation
Keywords: RenalTransplantation; KidneyTransplantation; MPA; EC-MPS
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Enteric-coated mycophenolate sodium (Experimental): Enteric-coated mycophenolate sodium tablets taken orally twice a day (in the morning and in the evening) at a dose equimolar to the dose of mycophenolate mofetil the participant was taking prior to start of the study + Placebo to mycophenolate mofetil capsules taken orally twice a day for 30 days. Participants remained on their standard immunosuppressive regimen of calcineurin inhibitors (CNI) (Cyclosporin A or Tacrolimus) administered with or without corticosteroids throughout the study.
  Interventions: Drug: Enteric-coated mycophenolate sodium (EC-MPS); Drug: Placebo to mycophenolate mofetil
- Mycophenolate mofetil (Active Comparator): Mycophenolate mofetil capsules taken orally twice a day (in the morning and in the evening) at the dose the participant was taking prior to study start + Placebo to mycophenolate sodium tablets taken twice a day for 30 days. Participants remained on their standard immunosuppressive regimen of calcineurin inhibitors (CNI) (Cyclosporin A or Tacrolimus) administered with or without corticosteroids throughout the study.
  Interventions: Drug: Mycophenolate mofetil; Drug: Placebo to mycophenolate sodium

INTERVENTIONS:
Drug: Enteric-coated mycophenolate sodium (EC-MPS) — Enteric-coated mycophenolate sodium supplied as 180 mg tablets.
  Other Names: Myfortic®
  Arms: Enteric-coated mycophenolate sodium
Drug: Mycophenolate mofetil — Mycophenolate mofetil supplied as 250 mg capsules.
  Arms: Mycophenolate mofetil
Drug: Placebo to mycophenolate sodium — Placebo to mycophenolate sodium matching tablets.
  Arms: Mycophenolate mofetil
Drug: Placebo to mycophenolate mofetil — Placebo to mycophenolate mofetil matching capsules.
  Arms: Enteric-coated mycophenolate sodium

SUMMARY:
Treatment with the immunosuppressive drug mycophenolate mofetil (MMF) may result in gastrointestinal (GI) complications in some patients. This study will investigate the safety and tolerability of converting kidney transplant recipients with gastrointestinal symptoms from their current treatment of mycophenolate mofetil (MMF) to treatment with enteric-coated mycophenolate sodium (EC-MPS).

ELIGIBILITY:
Inclusion criteria:

* Males and females aged 18-75 years, Recipients of first or second cadaveric, living unrelated or living related kidney transplant
* Recipients who are at least 4 weeks post renal transplantation with stable renal function, Patients currently receiving MMF (all dosages are allowed) and either cyclosporine USP (MODIFIED) or tacrolimus with or without corticosteroids as part of their immunosuppressive regimen for at least 2 weeks prior to study start
* Patients with at least one mild and/or moderate and/or severe upper or lower gastrointestinal (GI) complaints clearly associated with MMF therapy as determined by the treating physician. Additional mild GI complaints may coexist
* Patients' immunosuppressive regimen other than steroids (doses and type) as well as medication for treatment of GI symptoms must be unchanged for at least 1 week prior to study start
* Females of childbearing potential must have a negative pregnancy test prior to the inclusion period. The test should be performed locally at Baseline visit. If positive, the patient will not be included. Effective contraception must be used during the trial, and for 4 weeks following discontinuation of the study medication
* Patients who are willing and able to participate in the full course of the study and from whom written informed consent has been obtained.

Exclusion criteria:

* Multi-organ transplant patients (e.g. kidney and pancreas) or previous transplant with any other organ different from kidney (second kidney transplant is allowed)
* History of GI disorder (diarrhea, Gastroesophageal Reflux Disease (GERD), dyspepsia, Inflammatory Bowel Disease (IBD) or Irritable Bowel Syndrome (IBS) prior to transplantation
* Evidence of any GI disorder induced by an infection, underlying medical condition, or concomitant medication other than MMF, Modification of GI medication or MMF dose within last 1 week
* Evidence of graft rejection, treatment of acute rejection, or unstable renal function within 4 weeks prior to the Baseline visit, Patients who have received an investigational immunosuppressive drug within 4 weeks prior to study entry
* Patients with a history of malignancy within the last five years, except excised squamous or basal cell carcinoma of the skin
* Pregnant or nursing (lactating) women, Women of child-bearing potential (WOCBP) not using an acceptable method of contraception such as: surgical sterilization, hormonal contraception, or double-barrier methods.
* Contraception should be maintained throughout the study and for 4 weeks after study drug discontinuation.

Other protocol defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2006-10; Primary Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (53):
- United States (53):
  - AKDHC Medical Research Services, LLC, Phoenix, Arizona
  - University of Southern California, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - National Institute of Transplantation, Los Angeles, California
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - University of California San Diego, San Diego, California
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, California
  - Denver Nephrology, Denver, Colorado
  - University of Colorado Health Science Center, Denver, Colorado
  - Yale University Transplantation, New Haven, Connecticut
  - Washington Hospital Transplant Research, Washington D.C., District of Columbia
  - University of Florida College of Medicine, Gainesville, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Clarian Health Partners, Indianapolis, Indiana
  - Univ of KS Medical Ctr, Kansas City, Kansas
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Northwest Louisiana Nephrology Research, Shreveport, Louisiana
  - WKHS/LSUHSC Regional Transplant Center, Shreveport, Louisiana
  - University of Maryland, Baltimore, Maryland
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Mid-Atlantic Nephrology Associates, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - St. John Hospital Medical Center, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - St. Luke's Hospital of Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - St. Baranabas Medical Center, Livingston, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest, Winston-Salem, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Pinnacle Health at Harrisburg Hospital, Harrisburg, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - The University of Tennessee Health Science Center, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - CRSTI, Dallas, Texas
  - Baylor All Saints, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Utah Hospitals and Clinics, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Enteric-coated Mycophenolate Sodium | Mycophenolate Mofetil
Started | 200 | 200
Intent-to-Treat Population | 199 (Participants who received study drug.) | 197
Completed | 186 | 185
Not Completed | 14 | 15
Not completed — Adverse Event | 9 | 8
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Administrative Problem | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Did not receive study drug | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enteric-coated Mycophenolate Sodium | Mycophenolate Mofetil | Total
Number analyzed (Participants) | 199 | 197 | 396
Age Continuous [Mean (Standard Deviation); unit: Years] — Baseline Measures are based on the Intent-to-Treat (ITT) population that consisted of all randomized participants who received study drug.
  Years | 48.4 (13.4) | 48.4 (12.6) | 48.4 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 95 | 200
  Male | 94 | 102 | 196

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Who Responded to the Conversion to Mycophenolate Sodium (EC-MPS) Therapy
Description: Response assessed using the Gastrointestinal Symptom Rating Scale (GSRS), designed to assess common symptoms with gastrointestinal (GI) disorders. The GSRS has 5 subscales (reflux, diarrhea, constipation, abdominal pain and indigestion) producing a mean subscale score ranging from 1 (no discomfort) to 7 (very severe discomfort). The total score is an average of scores across all 15 items; a higher score indicates more GI symptoms. Response was defined as Day 30 improvement in the GSRS Total Score (change from baseline) of greater than or equal to 0.3. Minimum score is 1; maximum score is 7.
Time Frame: Baseline, Day 30
Population: Intention-to-treat (ITT) population consisted of all randomized participants who received at least one dose of study drug. 2 participants in the enteric-coated mycophenolate sodium group were excluded from the analysis because they had no baseline data.
Measure: Number; unit: Participants
Arm/Group | Enteric-coated Mycophenolate Sodium | Mycophenolate Mofetil
Number analyzed (Participants) | 197 | 197
Participants
  Response | 123 | 109
  No Response | 74 | 88

2. Secondary Outcome: Number of Participants With Biopsy-proven Acute Rejection (BPAR) and Treated Acute Rejection (TAR)
Description: TAR was defined as an episode of acute rejection that was suspected on clinical grounds and was treated and confirmed by the investigator according to the patient's response to therapy.
  BPAR was defined a treated acute rejection that was confirmed by biopsy. A graft core biopsy was performed before or within 24 hours of initiation of anti-rejection therapy and was assessed by the pathologist at the center according to the BANFF 1997 criteria.
Time Frame: 30 days
Population: Intent-to-treat population consisted of all randomized participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Enteric-coated Mycophenolate Sodium | Mycophenolate Mofetil
Number analyzed (Participants) | 199 | 197
Participants
  BPAR | 0 | 1
  TAR | 0 | 1

3. Secondary Outcome: Change From Baseline to Day 30 in the Severity of Gastrointestinal Symptoms Overall Total Score
Description: The Severity Score for each GI symptom for each participant was calculated based on the physician's evaluation of current GI symptoms recorded at Baseline and Day 30. For each of the 16 individual GI symptoms the severity score ranged from 0 (absent) to 3 (severe). The Overall Total Score is the Mean of severity ratings of the 16 individual symptoms.
Time Frame: Baseline, Day 30
Population: Intention to treat (ITT) population consisted of all randomized participants who received at least one dose of study drug. "n" in each of the categories is the number of participants with data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Enteric-coated Mycophenolate Sodium | Mycophenolate Mofetil
Number analyzed (Participants) | 199 | 197
Score on a scale
  Baseline (n= 198,195) | 0.7 (0.4) | 0.6 (0.4)
  Day 30 (n=193, 191) | 0.4 (0.4) | 0.4 (0.4)
  Change from Baseline to Day 30 (n=193,189) | -0.3 (0.4) | -0.2 (0.4)

4. Secondary Outcome: Number of Participants With Reported Dose Changes or Interruption of Study Medication During the 30 Days of Treatment
Description: The number of participants with reported dose changes or interruption of study medication during the 30 days of treatment.The most common dose adjustments were dose increases back to baseline levels following a decrease or interruption and decreases due to abnormal laboratory value Adverse Events (leucopenia, thrombocytopenia, neutropenia, or anemia).
Time Frame: 30 days
Population: Intention to treat (ITT) population consisted of all randomized participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Enteric-coated Mycophenolate Sodium | Mycophenolate Mofetil
Number analyzed (Participants) | 199 | 197
Participants
  Study drug change or interruption: YES | 11 | 12
  Study drug change or interruption: NO | 188 | 185

5. Secondary Outcome: Change From Baseline in Lower and Upper GI Symptom Burden Measured by GI Symptom Rating Scale Score
Description: This is reflected by the total score. The total score incorporates lower and upper GI elements. GSRS overall score is the mean of 15 individual GI symptom scores, each rated on a 7- point scale: 1 = no discomfort, 2= minor discomfort, 3 = mild discomfort, 4 = moderate discomfort, 5 = moderately sever discomfort, 6 = severe discomfort and 7 = very severe discomfort. Change from Baseline was calculated using ANCOVA, model includes GSRS, center and treatment group.
Time Frame: Baseline, Day 30
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Enteric-coated Mycophenolate Sodium | Mycophenolate Mofetil
Number analyzed (Participants) | 197 | 197
change in score on a scale | -0.6 (0.9) | -0.5 (1.0)

6. Secondary Outcome: Change in Gastrointestinal Symptom Rating Scale Subscale Scores After 30 Days of Treatment
Description: The GSRS has five subscales (reflux, diarrhea, constipation, abdominal pain, indigestion) producing a mean subscale score ranging from 1 (=no discomfort at all) to 7 (very severe discomfort). The mean score at baseline (BL), the mean score at Day 30 and the mean Change from BL to Day 30 is presented for each of the five subscales.
Time Frame: Baseline to Day 30
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Enteric-coated Mycophenolate Sodium | Mycophenolate Mofetil
Number analyzed (Participants) | 197 | 197
Score on a scale
  Diarrhea: Baseline (BL) | 3.3 (1.7) | 3.3 (1.7)
  Diarrhea: Day 30 | 2.4 (1.6) | 2.5 (1.6)
  Diarrhea: Change from BL to Day 30 | -0.9 (1.7) | -0.8 (1.6)
  Indigestion : Baseline | 2.8 (1.3) | 2.8 (1.3)
  Indigestion: Day 30 | 2.1 (1.0) | 2.4 (1.2)
  Indigestion: Change from BL to Day 30 | -0.7 (1.2) | -0.5 (1.4)
  Constipation: Baseline | 2.2 (1.2) | 2.1 (1.1)
  Constipation: Day 30 | 1.7 (0.9) | 1.8 (0.9)
  Constipation: Change from BL to Day 30 | -0.4 (1.1) | -0.3 (1.0)
  Abdominal pain: Baseline | 2.3 (1.1) | 2.5 (1.1)
  Abdominal pain: Day 30 | 1.8 (0.9) | 2.0 (1.1)
  Abdominal pain: Change from BL to Day 30 | -0.5 (1.1) | -0.5 (1.2)
  Reflux : Baseline | 2.2 (1.3) | 2.2 (1.4)
  Reflux : Day 30 | 1.7 (1.1) | 1.7 (1.1)
  Reflux : Change from BL o Day 30 | -0.5 (1.3) | -0.5 (1.5)

7. Secondary Outcome: Change From Baseline (BL) to Day 30 in the Gastrointestinal Quality of Life Index (GIQLI) Total Score and Subscale Scores
Description: The GIQLI is a 36-item questionnaire to assess the impact of GI disease on daily life. The GIQLI has 5 different subscales (GI symptoms, emotional status, physical and social functions, and stress of medical treatment) that are rated on a 5-point scale from 0 to 4. The individual scores are summed to produce a total score of the 36 items for a total possible score of 0 to 144. Lower scores represent greater dysfunction.
Time Frame: Baseline, Day 30
Population: Participants from the Intention-to-treat (ITT) population consisting of all randomized participants who received at least one dose of study drug for whom data was available for analysis. "n" in each of the categories is the number of participants with data available.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Enteric-coated Mycophenolate Sodium | Mycophenolate Mofetil
Number analyzed (Participants) | 197 | 197
Score on a scale
  Overall Total Score: BL ( n= 197,197) | 94.3 (17.9) | 93.4 (18.0)
  Overall Total Score : Day 30 (n= 195,192) | 105.0 (18.4) | 103.5 (18.1)
  Overall Total Score : Change from BL (n=193,192) | 10.7 (16.4) | 10.2 (17.5)
  GI Symptom: BL (n= 197, 197) | 46.7 (10.6) | 46.6 (10.3)
  GI Symptom: Day 30 (n= 195, 192) | 52.6 (10.8) | 51.9 (10.7)
  GI Symptom: Change from BL (n= 193, 192) | 5.9 (9.8) | 5.4 (10.2)
  Emotional Status: BL (n= 196, 197) | 11.9 (2.7) | 11.6 (2.9)
  Emotional Status: Day 30 (n= 195, 192) | 13.2 (2.8) | 13.1 (2.6)
  Emotional Status: Change from BL (n= 192, 192) | 1.3 (2.9) | 1.5 (3.0)
  Physical Function: BL (n= 196, 197) | 21.7 (3.8) | 21.5 (3.9)
  Physical Function: Day 30 (n= 195, 192) | 23.7 (3.4) | 23.3 (3.8)
  Physical Function: Change from BL (n= 192, 192) | 2.1 (3.2) | 1.9 (4.0)
  Social Function: BL (n= 197, 197) | 10.7 (2.8) | 10.4 (2.8)
  Social Function: Day 30 (n= 195, 192) | 11.9 (3.0) | 11.6 (2.8)
  Social Function: Change from BL (n= 193, 192) | 1.2 (2.6) | 1.2 (2.7)
  Medical treatment: BL (n= 197, 197) | 3.3 (1.0) | 3.4 (1.0)
  Medical treatment: Day 30 (n= 194, 192) | 3.6 (0.8) | 3.6 (0.7)
  Medical treatment: Change from BL (n= 192, 192) | 0.2 (1.0) | 0.3 (0.9)

ADVERSE EVENTS:
Arm/Group | Enteric-coated Mycophenolate Sodium | Mycophenolate Mofetil
Serious Adverse Events (participants affected / at risk) | 7/199 | 11/197
Other Adverse Events (participants affected / at risk) | 75/199 | 89/197
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enteric-coated Mycophenolate Sodium (N=199) | Mycophenolate Mofetil (N=197)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 2
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1 | 1
Weight decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lymphocele (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Enteric-coated Mycophenolate Sodium (N=199) | Mycophenolate Mofetil (N=197)
Abdominal distension (Gastrointestinal disorders) | 27 | 31
Abdominal pain lower (Gastrointestinal disorders) | 10 | 12
Abdominal pain upper (Gastrointestinal disorders) | 9 | 16
Constipation (Gastrointestinal disorders) | 7 | 15
Diarrhoea (Gastrointestinal disorders) | 21 | 17
Dyspepsia (Gastrointestinal disorders) | 19 | 17
Eructation (Gastrointestinal disorders) | 9 | 20
Flatulence (Gastrointestinal disorders) | 11 | 19
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 13 | 9
Intestinal functional disorder (Gastrointestinal disorders) | 10 | 14
Nausea (Gastrointestinal disorders) | 11 | 21
Decreased appetite (Metabolism and nutrition disorders) | 10 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.